CLINICAL TRIAL: NCT05462717
Title: Phase 1/1b, Multicenter, Open-Label, Dose Escalation and Dose Expansion Study of RMC-6291 Monotherapy in Subjects With Advanced KRASG12C Mutant Solid Tumors
Brief Title: Dose Escalation and Dose Expansion Study of RMC-6291 Monotherapy in Subjects With Advanced KRASG12C Mutant Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Revolution Medicines, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RMC-6291-001
Record Dates: First submitted 2022-07-11; First posted 2022-07-18 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-06

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC); Colorectal Cancer (CRC); Pancreatic Ductal Adenocarcinoma; Advanced Solid Tumor
Keywords: RMC-6291; RAS(ON); KRAS; KRASG12C; KRASG12C(ON); Targeted therapy; Metastatic cancer; Lung Cancer; Lung Neoplasms; Thoracic Neoplasms; Non-small Cell Lung Cancer; Carcinoma, Non-Small Cell Lung; NSCLC; Colorectal Cancer; Colonic Neoplasms; CRC; Appendiceal Cancer; KRAS mutation; STK11/LKB1; KEAP1; bronchial neoplasms; respiratory tract neoplasms; neoplasms by site; neoplasms; Colon Cancer; Rectal Cancer; lung disease; respiratory tract diseases; Pancreatic Cancer; Carcinoma, Pancreatic Ductal; PDAC; Gastrointestinal Neoplasms; Intestinal Neoplasms; Esophageal cancer; Ampullary cancer; Gastric Cancer; Gynecological Cancer; Ovarian Cancer; Endometrial Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Neoplasm Metastasis; Lung Neoplasms; Thoracic Neoplasms; Colonic Neoplasms; Appendiceal Neoplasms; Bronchial Neoplasms; Respiratory Tract Neoplasms; Neoplasms by Site; Neoplasms; Rectal Neoplasms; Lung Diseases; Respiratory Tract Diseases; Pancreatic Neoplasms; Carcinoma, Pancreatic Ductal; Gastrointestinal Neoplasms; Intestinal Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Ovarian Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RMC-6291 (Experimental): Dose Escalation and Dose Expansion
  Interventions: Drug: RMC-6291

INTERVENTIONS:
Drug: RMC-6291 — Oral tablet once or twice a day

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics (PK) of escalating doses of RMC-6291 (KRAS G12C(ON) inhibitor) monotherapy in adult subjects with advanced solid tumors and to identify the maximum tolerated dose (MTD), and the recommended Phase 2 dose.

DETAILED DESCRIPTION:
This is an open-label, multicenter, Phase 1/1b study of RMC-6291 monotherapy in subjects with advanced KRASG12C-mutant solid tumors. The study will include 2 components: a Dose-Escalation and a Dose-Expansion. Subjects will be treated until disease progression per RECIST v1.1, unacceptable toxicity, or other criteria for withdrawal are met, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be ≥18 years of age.
* Subject must have pathologically documented, locally advanced or metastatic KRASG12C-mutated solid tumor malignancy (not amenable to curative surgery) that has previously been treated with standard-of-care therapies for respective tumor types, is intolerant to, or is considered ineligible for standard-of-care anticancer treatments.
* ECOG performance status 0 or 1
* Prior treatment with a KRASG12C (OFF) inhibitor allowed for dose escalation
* Adequate organ function

Exclusion Criteria:

* Primary central nervous system (CNS) tumors
* Active brain metastases
* Known impairment of GI function that would alter the absorption
* Major surgical procedures within 28 days or non-study-related minor procedures within 7 days of treatment.
* Prior therapy with KRASG12C (ON) inhibitor

Other inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Estimated)
Dates: Start 2022-09-19 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events | up to 3 years
  Number of participants with adverse events
Dose Limiting Toxicities | The first 21 days (i.e. Cycle 1)
  Number of participants with dose limiting toxicities

SECONDARY OUTCOMES:
Maximum Observed Blood Concentration of RMC-6291 | 7 Cycles
  Cmax
Time to Reach Maximum Blood Concentration of RMC-6291 | 7 Cycles
  Tmax
Area Under Blood Concentration Time Curve of RMC-6291 | 7 Cycles
  AUC
Elimination Half-Life of RMC-6291 | 7 Cycles
  t1/2
Ratio of accumulation of RMC-6291 from a single dose to steady state with repeated dosing | 7 Cycles
  accumulation ratio
Overall Response Rate (ORR) | 3 years
  Overall response rate per RECIST v1.1
Duration of Response (DOR) | 3 years
  Duration of response per RECIST v1.1
Disease Control Rate (DCR) | 3 years
  Disease control rate per RECIST v1.1
Time to Response (TTR) | 3 years
  Time to response per RECIST v1.1
Progression-Free Survival (PFS) | 3 years
  Progression-free survival per RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Revolution Medicines, Inc., Study Director — Revolution Medicines, Inc.
Locations (64):
- United States (15):
  - Highlands Oncology Group, Springdale, Arkansas
  - UC Irvine Cancer Center, Orange, California
  - UC Davis Cancer Center, Sacramento, California
  - UCSF, San Francisco, California
  - University of Miami School of Medicine Sylvester Comprehensive Cancer Center, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - American Oncology Partners of Maryland, Bethesda, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - MSK Cancer Center, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - Tennessee Oncology, Nashville, Tennessee
  - Next Oncology, San Antonio, Texas
  - START, San Antonio, Texas
  - Next Oncology Virginia, Fairfax, Virginia
- Australia (4):
  - Southside Cancer Care Centre, Sydney, New South Wales
  - Peninsula & South Eastern Haematology and Oncology Group, Frankston, Victoria
  - Austin Health, Olivia Newton-John Cancer Research & Wellness Centre, Heidelberg, Victoria
  - South West Health Care, Warrnambool, Victoria
- Czechia (3):
  - NH Hospital a.s., Hořovice
  - Klinika onkologie a radioterapie, Fakultni Nemocnice Hradec Kralove, Hradec Králové
  - Onkologicka klinika, Fakultni Nemocnice Olomouc, Olomouc
- France (7):
  - ICO, Angers
  - CHU Bordeaux Hospital Saint-Andre, Bordeaux
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - CHU Nantes, Nantes
  - ICANS, Strasbourg
- Italy (6):
  - S.C. Oncologia Falck, Dipartimento Ematologia ed Oncologia Niguarda Cancer Center, Milan
  - Istituto Europeo Oncologico, Milan
  - Istituto Nazionale Tumori Fondazione G. Pascale, Napoli
  - Azienda Ospedaliero-Universitaria San Luigi Gonzaga, Orbassano
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Centro Ricerche Cliniche di Verona s.r.l., Verona
- Malaysia (2):
  - University Malaya Medical Centre, Kuala Lumpur
  - Sarawak General Hospital, Kuching
- Poland (3):
  - Instytut MSF Sp zoo, Lodz
  - Med - Polonia Sp. z o. o., Poznan
  - Narodowy Instytut Onkologii, Warsaw
- Serbia (3):
  - MSB General Hospital, Belgrade
  - Clinical hospital center Bezanijska Kosa, Belgrade
  - Institute for pulmonary diseases Sremska Kamenica, Kamenitz
- National Cancer centre Singapore, Singapore, Singapore
- South Korea (4):
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Korea University Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
- Spain (9):
  - NEXT Oncology IOB Hospital Quirónsalud, Barcelona
  - ICO Hospitalet, Barcelona
  - Clínica Universidad de Navarra, Madrid
  - MD Anderson Cancer Center, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Clinica Universidad de Navarra, Pamplona
  - Hospital Universitario Quirónsalud, Pozuelo de Alarcón
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario Miguel Servet, Zaragoza
- Taiwan (4):
  - E-DA hospital, Kaohsiung City, Yanchao District
  - Taipei Tzu Chi Hospital, New Taipei City
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
- Thailand (3):
  - Siriraj Hospital, Bangkok Noi
  - Chiang Mai University, Chiang Mai
  - Khon Kaen University, Khon Kaen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schulze CJ, Seamon KJ, Zhao Y, Yang YC, Cregg J, Kim D, Tomlinson A, Choy TJ, Wang Z, Sang B, Pourfarjam Y, Lucas J, Cuevas-Navarro A, Ayala-Santos C, Vides A, Li C, Marquez A, Zhong M, Vemulapalli V, Weller C, Gould A, Whalen DM, Salvador A, Milin A, Saldajeno-Concar M, Dinglasan N, Chen A, Evans J, Knox JE, Koltun ES, Singh M, Nichols R, Wildes D, Gill AL, Smith JAM, Lito P. Chemical remodeling of a cellular chaperone to target the active state of mutant KRAS. Science. 2023 Aug 18;381(6659):794-799. doi: 10.1126/science.adg9652. Epub 2023 Aug 17. PMID 37590355